## **Document Coversheet**

Study Title: U54 Pilot: Comparing Tobacco Product Susceptibility and Product Substitution by Relative Rurality and Alcohol Use

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 8/14/2025 |
| NCT Number: | NCT07010601 |
| IRB Number | 76582 |
| Coversheet created: | 9/15/2025 |

IRB Approval 8/14/2025 IRB # 76582 Exempt

Researchers in the Healthier Futures Lab at the University of Kentucky are inviting you to take part in this assessment. The primary purpose of this assessment is to measure decision-making related to money, different tobacco and alcohol commodities, and hypothetical purchasing behavior. The results of this survey may be published in peer-reviewed academic journals.

Your participation in this will require approximately 55 minutes answering surveys and completing the experimental tobacco marketplace. This study involves completing various decision-making tasks, questions related to tobacco use, and then directs to the "experimental market place" where you will have the opportunity to make hypothetical purchases for various tobacco products. The completion link for this study is at the end of the experimental tobacco marketplace.

You may not directly benefit from participation in this research, however your responses will help us understand decision making under certain conditions. Some volunteers experience satisfaction from knowing they have contributed to research that may possibly benefit others in the future.

Some information may be available to others (who submit a request) for tax reporting purposes. The researchers of this study will not attempt to connect your responses to your identity in any way. Prolific IDs will only be collected for the purposes of providing compensation.

If you decide to participate in this study, you are free to stop participating at any time. If you decide to stop participating after you begin the survey, you can leave early and still receive compensation by contacting us directly through Prolific or by emailing us at healthful@uky.edu. Please note that your compensation will be adjusted based on how much of the study you completed.

We may use the data we collect in this study in future research. Data will be deidentified before it is ever published and presented in aggregate form. Data used for analysis will be stored separately from your Worker ID and we will make no attempt to link your Worker ID with your answers.

We hope to receive completed questionnaires from about 800 people, so your answers are important to us. Of course, you have a choice about whether or not to complete the questionnaire. If you do participate, you are free to stop at any time. You will not be penalized in any way for discontinuing the survey. Please be aware that we make every effort to protect your data once received from the online survey company. Given the nature of online surveys, as with anything involving the internet, we can never guarantee the confidentiality of the data while still on the survey company's servers, or while data is being

transferred to either them or us. It is also possible the raw data collected for research purposes will be used for marketing or reporting purposes by the survey/data gathering company after the research is concluded, depending on the company's Terms of Service and Privacy policies.

Participating in this study will result in no risks greater than those which are found in everyday life. Answering questions related to substance use may be uncomfortable or embarrassing. If you would like more information about resources available to you for mental or substance use disorders, please visit:

https://www.samhsa.gov/findhelp/national-helpline.

If you have any questions about the study, please feel free to ask using the contact information below. Thank you in advance for your time and interest in participating in our research. If you have any questions or concerns about your rights as a research subject, you may contact the University of Kentucky Office of Research Integrity at (859) 257-9428 or toll-free at 1-866-400-9428.

Your consent to participate in this research is implied with submission of the assessment. If you do not choose to consent, please return this submission.

Sincerely, Mikhail Koffarnus, Ph.D.

College of Medicine,

University of Kentucky

Phone: 859-323-6402

Email: koffarnus@uky.edu